CLINICAL TRIAL: NCT07022041
Title: Sepsis Mortality in Hospitals: a Quality Indicator in Acute Care Settings
Brief Title: Sepsis and Hospital Mortality
Status: Recruiting | Type: Observational
Sponsor: University of Calabria (Other)
Responsible Party: Principal Investigator, Antonio Curcio, Professor, University of Calabria
Other Study IDs: 59/2025
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Electric Conductivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Sepsis
  Interventions: Diagnostic Test: conductivity and dieletric constant
- Myocarditis
  Interventions: Diagnostic Test: conductivity and dieletric constant
- Pericarditis
  Interventions: Diagnostic Test: conductivity and dieletric constant
- Endocarditis
  Interventions: Diagnostic Test: conductivity and dieletric constant
- Control Cases
  Interventions: Diagnostic Test: conductivity and dieletric constant

INTERVENTIONS:
Diagnostic Test: conductivity and dieletric constant — collecting blood samples and directly measuring plasma conductivity and dielectric constant using microwave probes already validated for non-invasive glucose monitoring.

SUMMARY:
Sepsis is one of the leading causes of hospital mortality, with a rate of approximately 20% (World Health Organization) among vulnerable patients admitted to high-intensity care units such as CCUs and inpatient wards. Currently, diagnostic criteria such as the Systemic Inflammatory Response Syndrome (SIRS) and the Sequential Organ Failure Assessment (SOFA) score, although widely used, lack sufficient specificity and accuracy. No established parameters are available for early and timely diagnosis. This study aims to address this gap by investigating the variability of blood plasma conductivity and dielectric constant using microwave probes previously validated for non-invasive glucose monitoring. The acquired data will be analyzed using the Anritsu VectorStar VNA to identify innovative and reliable parameters associated with the presence of severe infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cardiology patients without documented infection (Control Group)
* Patients with sepsis
* Patients with nosocomial infection
* Patients with myocarditis, endocarditis, or pericarditis
* Ability to provide written informed consent

Exclusion Criteria:

* Patients with severe or chronic medical conditions that may interfere with study results, such as autoimmune diseases, renal or hepatic failure
* Patients taking medications that could affect the measured biophysical parameters, such as corticosteroids or immunosuppressants
* Patients with cancer
* Patients with diseases involving the immune system (e.g., lymphomas, leukemias)
* Patients with congenital or acquired immunodeficiencies (e.g., HIV)
* Patients who are unable to read and sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cardiac patients aged 18 years and older, both with and without infections, are considered, while those with severe comorbidities or undergoing treatments that may influence the study outcomes are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Comparative Analysis of Plasma Bioelectrical Properties in Sepsis | through study completion, an average of 10 days
  differences in blood plasma conductivity and dielectric constant will be analyzed between patients with and without sepsis, using validated microwave probes and appropriate statistical methods.

SECONDARY OUTCOMES:
Correlation Between Biophysical Parameters and Conventional Infection and Inflammation Biomarkers | through study completion, an average of 3 months
  correlations will be assessed between measured biophysical parameters and conventional infection/inflammation biomarkers (e.g., ESR, procalcitonin, CRP, and white blood cell count) in patients with suspected or confirmed infection.

CONTACTS AND LOCATIONS:
Locations (1):
- ''Annunziata'' Hospital, Cosenza, Italy

IPD SHARING:
Plan to Share IPD: No